CLINICAL TRIAL: NCT07370766
Title: A Real-world, Longitudinal Observational Study of the Impact of Tildrakizumab on Patient Reported Outcomes in Patients With Moderate-to-severe Psoriasis in Canada
Brief Title: Impact of Tildrakizumab on Patient Reported Outcomes in Patients With Moderate-to-severe Psoriasis in Canada
Acronym: PRO/PsO
Status: Recruiting | Type: Observational
Sponsor: Chronicle Academy (Other)
Responsible Party: Sponsor
Other Study IDs: PRO/PsO-01
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis (PsO); Moderate to Severe Psoriasis
Keywords: psoriasis; moderate to severe psoriasis; Fitzpatrick scale; tildrakizumab; patient reported outcomes
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: all participants

SUMMARY:
This is a multi-centre, non-interventional, open-label, prospective observational study that will be conducted across Canada over 52-week duration. Approximately 80 patients who are initiating tildrakizumab as part of their routine care through the ILUMYA SUPPORT® Program and meet the study's eligibility criteria will be enrolled. Specifically, the study will enroll patients with Fitzpatrick scale skin types III and above.

The real-world impact, safety and effectiveness of tildrakizumab on patients with moderate-to-severe plaque psoriasis (PsO) remain largely undocumented in Canada, despite its approval in 2018. Given Canada's diverse population, this study presents an opportunity to evaluate tildrakizumab's quality of life, safety and effectiveness in specific demographic groups, particularly those patients with Fitzpatrick scale skin type III and above.

The findings from this study will help optimize care, address unmet needs, and ensure that treatment outcomes are inclusive and reflective of Canada's diverse population.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Diagnosis of moderate-to-severe chronic plaque-type PsO with Fitzpatrick scale type III or above (BSA >/=3%).
3. Candidate for phototherapy and/or systemic therapy.
4. Planning to initiate tildrakizumab as part of routine clinical care through the ILUMYA SUPPORT® Program for the treatment of plaque PsO but has not yet received their first dose.

   a. Decision to treat with tildrakizumab must be made independently of and prior to study recruitment.
5. Must be able to read, understand, and communicate in English.
6. Must be willing to participate in the study and capable to provide informed consent
7. Able to comply with all study procedures and attend all study visits

Exclusion Criteria:

1. Known hypersensitivity to tildrakizumab, its excipients, or components of the container, as outlined in the Product Monograph.
2. Concurrently taking any oral medication for treatment of PsO (e.g. methotrexate, cyclosporin, acitretin)
3. Diagnosis of only palmoplantar psoriasis
4. Concurrent medical condition or significant comorbidities that, in the investigator's opinion, would prevent participation in the study or interfere with study assessments
5. Women of childbearing potential who are pregnant, planning to become pregnant, or breastfeeding.
6. Prior (within 30 days) or actively participating in other interventional clinical trial(s).
7. Unable or unwilling to comply with study procedures including completing questionnaire.
8. Any other condition that, in the opinion of the investigator, could create a hazard to the participant's safety, endanger the study procedures, or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate-to-severe psoriasis (PsO) planning to initiate treatment with tildrakizumab and meet Fitzpatrick scale skin type III or above.
  Patients that are either naïve to PsO treatment with a biologic or those who have previously been exposed to a biologic PsO treatment will be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of tildrakizumab on the Dermatology Life Quality Index (DLQI and DLQI-R) in patients of Fitzpatrick skin type III and above to 16 weeks | 16 weeks
  DLQI consists of 10 items designed to assess multiple domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Patients respond to each item based on their experiences over the past week, using a four-point scale that ranges from: 0 (not at all or not relevant), 1 (a little), 2 (a lot), 3 (very much). Total DLQI score is calculated by summing the scores for all 10 items, resulting in a possible range from 0 to 30, where higher scores indicate greater impairment in QoL due to the skin condition. DLQI-Relevant adjusted for non-relevant answers

SECONDARY OUTCOMES:
Evaluate the impact of tildrakizumab on DLQI and DLQI-R in patients of Fitzpatrick skin type III and above to 52 weeks | 52 weeks
  Evaluated using DLQI questionnaire; DLQI-Relevant adjusted for non-relevant answers
Evaluate efficacy of tildrakizumab using Psoriasis Area Severity Index (PASI) in patients with Fitzpatrick skin types III and above | Week 16, Week 52
  Absolute and percent change from baseline to Week 16 and 52. Number and percent of patients achieving PASI 75, PASI 90, PASI 100 at Week 16 and 52
Evaluate efficacy of tildrakizumab using Body Surface Area (BSA) in patients with Fitzpatrick skin types III and above | Week 16, Week 52
  Absolute and percent change from baseline to Week 16 and 52
Evaluate efficacy of tildrakizumab using static Physician Global Assessment (sPGA) in patients with Fitzpatrick skin types III and above | Week 16, Week 52
  Absolute and percent change from baseline to Week 16 and 52. Number and percent of participants achieving score 0 or 1 with at least a 2-grade reduction from baseline at Week 16 and 52
Impact of tildrakizumab treatment on quality of life | Week 16, Week 52
  Measured using Skindex-16 patient questionnaire. It consists of 16 items that assess three key domains affected by skin disease: symptoms, emotional impact, and functioning. Patients are asked to rate how often they experienced various impacts from their skin condition over the last seven days, using a seven-point response scale (0-6) that ranges from: 0 (never bothered) to 6 (always bothered). Absolute and percent change from baseline to Week 16 and 52 are calculated.
Impact of tildrakizumab treatment on sleep | Week 16, Week 52
  Measured using Medical Outcomes Study Sleep Scale (MOS-Sleep) patient questionnaire. Absolute and percent change from baseline to Week 16 and 52. Consisting of 12 items, MOS-Sleep measures subjective experiences of sleep across several different domains. Question 1 is a numerical scale 1-5, where 5 indicates most difficulty to fall asleep; question 2 asks average number of hours slept per night in last 4 weeks; questions 3-12 are numerical scale 1-6, where 1 is "all of the time" and 6 is "none of the time".
Impact of tildrakizumab treatment on discomfort | Week 16, Week 52
  Measured using Worst Itch Numerical Rating Scale (WI-NRS). Participants will use the NRS to rate their itch and skin pain, separately, on a scale ranging from 0 to 10, where: 0 indicates no skin pain or no itch, and 10 indicates the worst imaginable pain or itch. A 24-hour recall period will be applied.
  Absolute and percent change from baseline to Week 16 and 52 are calculated.
Impact of tildrakizumab on skin pain | Week 16, Week 52
  Measured using Skin Pain Numerical Rating Scale (SP-NRS) . Participants will use the NRS to rate their itch and skin pain, separately, on a scale ranging from 0 to 10, where: 0 indicates no skin pain or no itch, and 10 indicates the worst imaginable pain or itch. A 24-hour recall period will be applied.
  Absolute and percent change from baseline to Week 16 and Week 52 are calculated.
Evaluate the correlation between clinical improvement (PASI, BSA, sPGA) and QoL outcomes, identifying how improvements in disease severity align with enhancements in QoL measures. | Week 16, Week 52
  Change from baseline to Week 16 and 52 on PASI, BSA, sPGA vs. Change from baseline at Week 16 and 52 on DLQI, DLQI-R, Skindex-16, and MOS-Sleep
Evaluate the safety of tildrakizumab over the course of the study | Baseline to Week 52
  Number and percent of treatment emergent Adverse Events and Serious Adverse Events over time. Number of events of unusual failure in efficacy over course of study.
Assess patient adherence and satisfaction with tildrakizumab treatment | Baseline to Week 52
  Treatment satisfaction questionnaire for medication (TSQM-9) score at Week 16 and 52. The TSQM-9 measures satisfaction across four key domains: a) Effectiveness: How well the treatment controls symptoms b) Side Effects: The patient's experience of side effects, if any, c) Convenience: How easy it is to use the treatment, d) Global Satisfaction: The overall satisfaction with the medication. Participants will rate individual items using a 7-point Likert scale ranging from "Extremely Dissatisfied" to "Extremely Satisfied." Number and type of participant withdrawals. Number of missed tildrakizumab treatments (self-report)

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Burlington Skin and Wellness, Burlington, Ontario
  - Locke Dermatology, Hamilton, Ontario
  - Panorama Dermatology Clinic, Kanata, Ontario
  - Centricity Research London Victoria Multispecialty, London, Ontario
  - Factor Dermatology, Ottawa, Ontario
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No